CLINICAL TRIAL: NCT01838109
Title: Multicenter, Prospective Randomized Controlled Trial Evaluating Postoperative Oral Nutritional Supplementation for the Patients Who Received Major Gastrointestinal Surgery
Brief Title: Postoperative Oral Nutritional Supplementation After Major Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSSMN-01
Record Dates: First submitted 2013-04-10; First posted 2013-04-23 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2013-09

CONDITIONS: Gastric Cancer; Colon Cancer; Pancreatic Cancer; Duodenal Cancer; Biliary Cancer; Peptic Ulcer; Inflammatory Bowel Diseases
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Duodenal Neoplasms; Biliary Tract Neoplasms; Peptic Ulcer; Inflammatory Bowel Diseases | interventions — Dietary Supplements

ARMS (2):
- ONS group (Experimental): oral administration of Encover 2 package for day starting at the time of discharge (200ml/package x 2, total 400Kcal/day) total 87 patients
  Interventions: Dietary Supplement: oral nutritional supplement
- Control group (No Intervention): no intervention total 87 patients

INTERVENTIONS:
Dietary Supplement: oral nutritional supplement
  Other Names: Encover
  Arms: ONS group

SUMMARY:
Patients who underwent major gastrointestinal surgery is potentially at risk of malnutrition due to reduced oral intake, increased nutritional need, reduced gastrointestinal absorption function, and/or metabolic changes after surgery. The postoperative malnutrition is associated with low quality of life and seems to be related long-term nutritional status. This study is a multicenter, open-labeled prospective randomized clinical trial to examine the effect of postoperative oral nutritional supplements (ONS) after major gastrointestinal surgery by comparing the change of body weight and other nutritional parameters between the experiment group that is supplied with ONS and the control group without ONS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who are 20 or more years old and not more than 80 years old
* Discharge from a hospital is planned within 2 weeks after major gastrointestinal surgery (except when ileostomy is performed)
* oral intake is possible at the time of discharge
* no preoperative chemotherapy or preoperative radiotherapy
* voluntarily agreed with the informed consent of this clinical trial

Exclusion Criteria:

* Intravenous or other specific nutritional treatment is needed
* BMI >25 and postoperative weight loss is not > 5% of preoperative body weight at the time of discharge
* Allergy to milk, whey, bean, salmon, or the investigational product
* Residual of cancer in the abdominal cavity postoperatively if it is cancer case
* Presence of synchronous other cancers that needs treatment.
* When investigator judged that the patient is not eligible to the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Body weight decrease rate 8weeks after discharge compared with preoperative body weight | 8weeks after discharge

SECONDARY OUTCOMES:
Changes in body weight before and after surgery | preoperatively, at the time of discharge, and 2,4, 8 weeks after discharge
Change of body mass index before and after surgery | preoperatively, at the time of discharge after surgery, and 8 weeks after discharge
changes in PG-SGA score and grade | preoperatively, and 2,4,8 weeks after discharge
serum hemoglobin | preoperatively, at the time of discharge, 2,4,8 weeks after discharge
serum total lymphocyte count | preoperatively, at the time of discharge, 2,4,8 weeks after discharge
serum total cholesterol | preoperatively, at the time of discharge, 2,4,8 weeks after discharge
serum total protein | preoperatively, at the time of discharge, 2,4,8 weeks after discharge
serum albumin | preoperatively, at the time of discharge, 2,4,8 weeks after discharge

OTHER OUTCOMES:
Anthropometric measure (Triceps Skinfold Thickness and Mid Arm Muscle Circumference), optional | pre-operatively, and 2,4,8 weeks after discharge
ONS related gastrointestinal adverse event | upto 8weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Joon Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea